CLINICAL TRIAL: NCT07114289
Title: Comparison of Pressure Support Ventilation and T-Piece as Spontaneous Breathing Trials Before Extubation Among Obese and Overweight Patients
Brief Title: Spontaneous Breathing Trials Using Pressure Support or T-Piece in Overweight and Obese Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: N202412012
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-05

CONDITIONS: Mechanical Ventilation; Extubation; Obesity &Amp; Overweight; Respiratory Failure
MeSH Terms: conditions — Obesity; Overweight; Respiratory Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSV group (Active Comparator)
  Interventions: Procedure: Spontaneous breathing trial using pressure support ventilation
- T-Piece group (Active Comparator)
  Interventions: Procedure: Spontaneous breathing trial using T-Piece

INTERVENTIONS:
Procedure: Spontaneous breathing trial using pressure support ventilation — Patients will receive low level pressure support ventilation for 1 hour before extubation
  Arms: PSV group
Procedure: Spontaneous breathing trial using T-Piece — Patients will receive a T-piece with oxygen for 1 hour before extubation
  Arms: T-Piece group

SUMMARY:
This study aims to find out which method of spontaneous breathing trial (SBT) better helps overweight and obese ICU patients prepare for extubation, which is the removal of the breathing tube. The two methods being compared are pressure support ventilation (PSV) and the T-piece.

Participants are adults with a body mass index (BMI) of 25 or higher who have been on a breathing machine (invasive mechanical ventilation) for more than 24 hours. Before removing the breathing tube, participants will be randomly assigned to receive either a PSV or a T-piece trial for 1 hour. After that, doctors will decide if they are ready for extubation.

The main question this study wants to answer is: Which method leads to a higher rate of successful extubation-defined as not needing to be reintubated within 72 hours?

ELIGIBILITY:
Inclusion Criteria:

1. Patients had undergone intubation and mechanical ventilation for more than 24 hours prior to the first spontaneous breathing trial.

2. Adult patients aged ≥ 18 years. 3. BMI ≥ 25 kg/m². 4. Meeting all the Inter national Consensus Conference on weaning criteria:

1. Stable vital signs: heart rate < 140 beats/min, systolic blood pressure: 90-160 mmHg, and no use of vasopressors or use of minimal doses (<0.2 µg/kg per min).
2. Respiratory rate ≤ 35 breaths/min.
3. Adequate oxygenation, defined as either SpO2 > 90% with FiO2 ≤ 0.4, or PaO2/FiO2 > 150 mmHg with positive end-expiratory pressure (PEEP) ≤ 8 cmH2O.
4. Adequate cough strength (MIP < -20 cmH2O).
5. An awake state, defined as a score of Richmond Agitation-Sedation Scale between +1 and -2, or Glasgow Coma Scale > 8.
6. No continuous sedation. 5. Informed consent provided by the patient or their relatives.

Exclusion Criteria:

1. Patients with tracheostomy.
2. Patients who had been admitted for traumatic brain injury.
3. Patients who had preexisting peripheral neuromuscular disease (underlying myopathy or myasthenia gravis).
4. Patients who had a do-not-reintubate order at the time of the initial spontaneous breathing trial were excluded
5. Patients who have already undergone a first spontaneous breathing trial.
6. Patients who had undergone extubation without an SBT
7. Protected populations: pregnant or breastfeeding women, individuals under guardianship, or those under legal protection.
8. Patients who refused to participate during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Successful extubation within 72 hours | Within 72 hours after extubation

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan